CLINICAL TRIAL: NCT04097899
Title: Impact of Implementation of Antimicrobial Stewardship Comprehensive Care Bundle Program on Ventilator Associated Pneumonia in Surgical Intensive Care Unit
Brief Title: Antimicrobial Stewardship Program and Ventilator Associated Pneumonia
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Michael Adel Shaker, lecturer of anesthesia, Zagazig University
Other Study IDs: 2143/11-5-2015
Record Dates: First submitted 2019-08-31; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — sputum culture and sensitivity
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A in preimplementation phase: Patient and antibiotic related data were collected to calculate and define; ventilator associated pneumonia incidence, mean ventilation days and mean length of stay, antibiotic selection, antibiotic cost, antibiotic susceptibility pattern, antibiotic consumption.
- Group B in postimplementation phase: The appropriateness of antibiotic use (selection, initiation, duration & time of discontinuation) before and after implementing the educational program was compared, calculation of the change in the ventilator associated pneumonia incidence & length of ICU stay, calculation of the change in the rate of antibiotic resistance and calculation of the cost change of antibiotics used after implementing the educational program.
  Interventions: Other: implementation of antimicrobial stewardship comprehensive care bundle program on ventilator associated pneumonia patients

INTERVENTIONS:
Other: implementation of antimicrobial stewardship comprehensive care bundle program on ventilator associated pneumonia patients — Construction of a comprehensive care bundle educational program. This program consisted of many elements: Antimicrobial stewardship programs, VAP bundles and infection control policy implementation and the investigators studied the impact of this program on:
  * Antibiotics cost.
  * Appropriates of antibiotic use (initiation, duration & time of discontinuation).
  * Rate of resistance
  * Clinical outcome, infection rate &length of stay.
  Groups: Group B in postimplementation phase

SUMMARY:
Antibiotic Stewardship Programs (ASPs) help clinicians improve the quality of patient care and improve patient safety through increased infection cure rates, reduced treatment failures; however, there are different techniques, with variable results, of its application including what is called ASPs bundle and there is a need to investigate the effectiveness of implementing a comprehensive care bundle program including the key components of ASPs and the key items of infection control measures, this program can be called Antimicrobial Stewardship Comprehensive Care Bundle Program (ASCCBP).

DETAILED DESCRIPTION:
Survey experimental study will be done in the first 6 months as regard antimicrobial drugs pattern and organism's sensitivity and resistance pattern in VAP patients.

In the next six months, clinical implementation of ASPs and infection control bundle will be applied on VAP patients. Then, in the later six months the investigators will study the outcome of VAP patients as regard:

* Amount of cost of antibiotics.
* Appropriates of antibiotic use (initiation, duration & time of discontinuation).
* Rate of resistance
* Clinical outcome, infection rate &length of stay.

Regular reports on antibiotic use and resistance will be admitted to relevant staff every one month. Also, audit and feedback about resistance and optimal prescribing will be applied every one month for ICU stuff as an open discussion.

The stewardship consulting team will include microbiologist with clinical experience in the field of antibiotic use and infection control. Stewardship team also will include the relevant ICU staff and an experienced clinical pharmacist.

ELIGIBILITY:
Inclusion Criteria:

• Patients, ≥18 years, who were intubated and mechanically ventilated for more than 48 hours in ICU and showing clinical criteria of VAP

Exclusion Criteria:

* Patients on immunosuppressive drugs.
* Patient with chronic lung disease, chronic liver disease& chronic renal disease.
* Immunocompromised Patients.
* Patients intubated and mechanical ventilated outside the ICU before admission.
* Patients manifested clinically with picture suggestive of VAP but less than 48 hours on mechanical ventilation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, ≥18 years, who were intubated and mechanically ventilated for more than 48 hours in ICU and showing clinical criteria of VAP. Diagnosis was based on the clinical pulmonary infection score then it was confirmed microbiologically by culture results. Clinical VAP criteria included the presence of a new or progressive pulmonary infiltrates on chest radiograph, fever (greater than 38.3°C), leukocytosis or leucopenia and appearance of purulent tracheobronchial secretions
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
change in ventilator associated pneumonia incidence | 18 months
  After implementation of the Antimicrobial Stewardship Comprehensive Care Bundle Program (ASCCBP), the percentage of VAP incidence was measured to assess the effectiveness of the program.
change in antibiotic resistance pattern | 18 months
  measuring the change in sensitivity and resistance pattern of antibiotics used in ICU was done by assessing the change in the sputum culture and sensitivity results.

SECONDARY OUTCOMES:
ventilation days | 18 months
  Days of mechanical ventilation of each patient were measured to calculate the difference before and after implementation of the program.
antibiotic cost | 18 months
  costs of antibiotics by Egyptian pounds were calculated to assess the effectiveness of the program

CONTACTS AND LOCATIONS:
Overall Officials: michael shaker, MD, Principal Investigator — faculty of medicine, Helwan university, Egypt; Heba Matar, MD, Study Director — faculty of medicine, zagazig university, Egypt; sahar saad-eldeen, MD, Study Director — faculty of medicine, zagazig university, Egypt; Rehab elsokkary, MD, Study Director — faculty of medicine, zagazig university, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data could be shared
Supporting Information: Study Protocol
Time Frame: indefinite time
Access Criteria: Easy, direct information are available for other researchers